CLINICAL TRIAL: NCT04031040
Title: A Post-market Clinical Follow up of the Genio® System for the Treatment of Obstructive Sleep Apnea in Adults.
Acronym: EliSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nyxoah S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-GEN-002068
Record Dates: First submitted 2019-07-18; First posted 2019-07-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genio® system therapy (Experimental): Following activation of the Genio® system at 8 weeks post-surgery, patients will be followed at 12 weeks, 6 months, 9 months, 12 months and then every year for a total period of 5 years after surgery.
  Interventions: Device: Genio® system therapy

INTERVENTIONS:
Device: Genio® system therapy — Hypoglossal nerve stimulation system

SUMMARY:
The primary objective of this study is to confirm the safety and clinical effectiveness of the Genio® system in moderate to severe Obstructive Sleep Apnea (OSA) adult patients over a period of 5 years post-surgery.

DETAILED DESCRIPTION:
This study is a multicenter, prospective single arm PMCF. Following activation of the Genio® system between 6 to 10 weeks post-surgery, patients will be followed at 3 months, 6 months, 9 months, 12 months and then every year for a total period of 5 years after surgery. Phone calls follow-up will be performed at Month 18, Month 30, Month 42 and Month 54.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) < 35 kg/m2
* AHI between 15 to 65 events/hour documented by the closest PSG performed at the time of the patient ICF signature and within maximum 12 months of screening and fulfilling the required technical criteria or during the screening phase.
* Has either not tolerated, has failed or refused Positive Airway Pressure (PAP) or Mandibular Advancement Device (MAD) treatments.

Exclusion Criteria:

* Inadequately treated sleep disorders other than OSA that would confound functional sleep assessment;
* Taking medication that in the opinion of the Investigator may alter consciousness, the pattern of respiration, or sleep architecture;
* Major anatomical or functional abnormalities that would impair the ability of the Genio® system to treat OSA;
* Inadequately treated psychiatric disease that prevent patient compliance with the requirements of the investigational study testing;
* Life expectancy < 12 months;
* Participation in another clinical study (excluding registries) during the study period (3 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of device-related Serious Adverse Events (SADEs) | 12 months post-surgery
  Incidence of device-related Serious Adverse Events (SADEs)
Change in Apnea-Hypopnea Index from baseline | 12 months post-surgery
  Change in Apnea-Hypopnea Index (AHI) from baseline as measured by sleep lab
Change in the quality of life measured by the Functional Outcomes of Sleep Questionnaire | 12 months post-surgery
  Change in the quality of life measured by the Functional Outcomes of Sleep Questionnaire (FOSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim T. Maurer, MD, Principal Investigator — Klinik für HNO-Heilkunde, Mannheim
Locations (21):
- Belgium (2):
  - Ziekenhuis Netwerk Antwerpen - ZNA Jan Palfijn, Antwerp
  - Universitair Ziekenhuis Antwerpen, Antwerp
- France (12):
  - CHU - Angers, Angers
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Henri-Mondor AP-HP, Créteil
  - Hôpital Privé La Louvière, Lille
  - Clinique Beau-Soleil, Montpellier
  - Hôpital Bichat, Assistance Publique - Hôpitaux de Paris, Paris
  - CEREVES Paris Jean Jaurès - Centre du sommeil, Paris
  - Hôpital Tenon AP-HP, Paris
  - CHU - Poitiers, Poitiers
  - Clinique Mutualiste de la Sagesse, Rennes
  - Polyclinique Saint Laurent, Rennes
  - CHU Toulouse, Toulouse
- Germany (5):
  - Asklepios Klinikum Harburg, Abt. für HNO-Heilkunde, Kopf- und Halschirurgie, Hamburg
  - HNO-Klinik des Universitätsklinikums Jena, Jena
  - Klinik für HNO-Heilkunde, Kopf- und Halschirurgie, Schlafmedizinisches Zentrum, Mannheim
  - Klinikum rechts der Isar der TU München, München
  - Helios Universitätsklinikum Wuppertal,Klinik für Hals-Nasen-Ohrenheilkunde, Kopf- und Halschirurgie, Wuppertal
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands
- Kantonsspital Baselland, Klinik für HNO-Krankheiten, Kopf- und Gesichtschirurgie, Liestal, Switzerland